CLINICAL TRIAL: NCT03160950
Title: Evaluating the Longevity and Safety of Full-coverage Crowns Fabricated With LuxaCrown Over a Period of 5 Years in 25-60 Year Old Indian Population: An Uncontrolled Trial
Brief Title: Clinical Efficacy of Crowns Fabricated Using LuxaCrown
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DMG Dental Material Gesellschaft mbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEPEND
Record Dates: First submitted 2017-05-15; First posted 2017-05-19 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: LuxaCrown; Single Crown Restoration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LuxaCrown (Experimental)
  Interventions: Device: LuxaCrown

INTERVENTIONS:
Device: LuxaCrown — Teeth that would be requiring RCT, would be initially treated by a endodontist using the standardized principles of rotary endodontics.
  Restoration using the LuxaCrown as a direct composite crown: In short, the impression material will be loaded with the LuxaCrown material (DMG, Germany). Approx. 0:40 minutes after the start of mixing, the filled impression will be placed in the patient's mouth and will stay there for approx. 1:45 - 2:20 minutes, that is, till the material is partially set. The impression will then be taken out and the material will be allowed to set outside patient's mouth up to approximately 5 minutes after the start of mixing. The Crown will then be finished using a fine buff and pumice, followed by application of Glaze and Bond (DMG, Germany). The preparation will then be cleaned and slightly roughened with a bur or sand blaster at the adhesion sites. The crown fabricated will then be cemented using PermaCem 2.0 luting cement (DMG, Germany).

SUMMARY:
A single arm non-blinded study is planned to evaluate the durability of the crowns fabricated using a novel composite based material, LuxaCrown (DMG, Germany). The durability of these crowns will be assessed for anatomical form, marginal adaptation, color match, marginal discoloration, surface roughness, secondary caries, pulpal compatibility, plaque index and modified papillary bleeding index with intensive follow up for 2 years (at 1 week, 3rd, 6th, 12th, 18th and 24th month), and then a yearly follow-up for additional 3 years (at 36th, 48th and 60th month).

A total of 50 patients will be selected and one tooth per subject will be included. For the purpose of study only the healthy adult patients with age range of 25 - 60 years who would be requiring Single crown restoration in the permanent anterior / posterior teeth, either due to caries, pulpal involvement or trauma, will be selected. Teeth that require endodontic treatment shall be included in the study only after successful endodontic therapy has been completed by an experienced endodontist. For broken teeth, only the teeth with > 1/2 crown structure remaining or in case of teeth with <1/2 crown structure fractured that can be restored with conventional post and core will be selected. In general, patients with bruxism, or with severe periodontal disease, mobility grade 2 or 3 shall be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patients with age range 25 - 60 years
* Only the patients who would be requiring Single crown restoration in the permanent anterior / posterior teeth will be selected for the purpose of study. Single crowns are usually indicated in either of the following conditions

  * Extensive coronal / structural broken tooth due to caries or trauma
  * Teeth undergone successful endodontic therapy (no signs of failure- asymptomatic, no tenderness on percussion, healthy associated soft tissue)
  * Microdonts

Teeth that require endodontic treatment shall be included in the study only after successful endodontic therapy has been completed by an experienced endodontist. The success of the endodontic therapy shall be evaluated using the standardized clinical and radiographic criteria by the endodontist.

* Broken teeth with > ½ crown structure remaining will be selected.
* Broken teeth with < ½ crown structure remaining will also be selected provided they can be restored with a crown after a conventional Post and core.
* Patients with good Occlusal Contact will be selected.
* Patients who would be giving the Signed Informed Consent shall only be enrolled for the study.
* Only the teeth showing mobility grade 0 and 1 as per Miller's Criteria shall be selected for the purpose of study.

Exclusion Criteria:

* Patients showing signs of bruxism shall not be selected. History of bruxism and wear facets will be checked for ruling out the bruxism habit.
* Patients with severe periodontal disease, that involves all teeth or tooth indicated for crown fabrication shall not be included in the study.
* Any clinical or radiographic sig or symptom indicative of periapical or furcation involvement.
* If the tooth indicated for crown fabrication depicts a mobility grade 2 or 3 as per Miller's criteria, it shall be excluded from the study.
* History of any systemic illness, pregnancy or history of allergy to dental fillings/materials shall also be excluded.
* Teeth with fracture of crown en-masse (Ellis Class VIII) fracture or which are badly mutilated such that a very minimal or No coronal structure is remaining will be excluded.
* Hypoplastic / malformed teeth will not be selected for the purpose of study.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change of anatomical form | 1 week, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Anatomical form will be assessed and scored according to Dijken modification of USPHS criteria.
Change of marginal adaptation | 1 week, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Marginal adaptation will be assessed and scored according to Dijken modification of USPHS criteria.
Change of color match | 1 week, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Color match will be assessed and scored according to Dijken modification of USPHS criteria.
Change of marginal discoloration | 1 week, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Marginal discoloration will be assessed and scored according to Dijken modification of USPHS criteria.
Change of surface roughness | 1 week, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Surface roughness will be assessed and scored according to Dijken modification of USPHS criteria.
Change of secondary caries | 1 week, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Secondary caries will be assessed and scored according to Dijken modification of USPHS criteria.
Change of wear | 1 week, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  The severity of attrition will be scored as described by Pergamalian
Change of pulpal compatibility | 1 week, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Assessment of the pulpal response by the FDI criteria
Change of plaque index | 1 week, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Plaque index will be assessed and scored according to Sillness and Loe, 1964
Change of modified papillary bleeding index | 1 week, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Measurement and scoring of modified papillary bleeding index (Barnett et al.)

SECONDARY OUTCOMES:
Change of patient satisfaction | 1 week, 3 months, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Patient satisfaction will be assessed by FDI criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Gugnani, Dr., Principal Investigator — Department of Pedodontics and Preventive Dentistry, DAV Dental College
Locations (1):
- DAV (C) Dental College Model Town, Yamuna Nagar, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided